CLINICAL TRIAL: NCT02644122
Title: A Phase II Open Label Study of the PI3 Kinase (PI-3) Inhibitor, SF1126, in Patients With Recurrent or Progressive SCCHN and Mutations in PIK3CA Gene and/or PI-3 Kinase Pathway Genes
Brief Title: SF1126 in Recurrent or Progressive SCCHN and Mutations in PIK3CA Gene and/or PI-3 Kinase Pathway Genes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Ezra Cohen (Other)
Collaborators: SignalRX Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ezra Cohen, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140904
Record Dates: First submitted 2015-12-07; First posted 2015-12-31 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma
Keywords: advanced cancer; metastatic cancer; Squamous Cell Carcinoma of the Head and Neck; SCCHN; gene mutation; PIK3R1, PIK3R5 and PIK3AP1; PIK3CG; AKT and mTOR; PIK3CA gene; PI-3 kinase inhibitor; PI-3 kinase pathway genes
MeSH Terms: conditions — Neoplasm Metastasis; Squamous Cell Carcinoma of Head and Neck; Hereditary Sensory and Autonomic Neuropathies | interventions — SF 1126

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SF1126 (Experimental): SF1126 1110 mg/m2 administered intravenously (IV) twice per week (separated by at least three days) for the first four treatment cycles (28 days) and then once weekly for subsequent cycles.
  Interventions: Drug: SF1126

INTERVENTIONS:
Drug: SF1126

SUMMARY:
The purpose of this study is to test the good and bad effects of an experimental drug called SF1126. This drug is being tested in patients whose cancer has not been controlled by available standard therapies and who have certain genes in their tumor.

SF1126 is a drug that inhibits a cell protein called phosphatidyl inositol 3 kinase (PI3K). PI3K is part of signaling pathway that tells cancer cells to grow, survive, invade and metastasize. PI3K also has an important role in the development of blood vessels that are required to support tumor growth. SF1126 is being developed by SignalRx Pharmaceuticals, Inc. It is considered an experimental drug because it is not approved by the FDA for any disease treatment.

DETAILED DESCRIPTION:
SignalRx Pharmaceuticals has developed a pan isoform specific PI-3 inhibitor called SF1126 to treat patients with advanced or metastatic cancer. SF1126 is a conjugate that contains two components: SF1101 (the active drug) and SF1174 (an inactive tetrapeptide RGD targeting moiety)

Both components of SF1126 play key roles in the activity of the drug. SF1101 is a selective inhibitor of certain members of the phosphatidyl inositol 3-kinase (PI-3) family and SF1174 binds selectively to receptors known to be present on neovasculature supporting tumors and on some tumor cells themselves. These components result in a drug designed to be both selective in its activity and targeted in its delivery.

This is an open label Phase II study of SF1126 in adult patients with recurrent or refractory advanced SCCHN with PIK3CA mutation. Treatment cycles (28 days) will consist of SF1126 1110 mg/m2 administered intravenously (IV) twice per week (separated by at least three days) for the first four cycles and then once weekly for subsequent cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent or metastatic SCCHN or any site except lip, thyroid, salivary gland, or nasopharynx.
* No known FDA-approved therapy available that's expected to prolong survival by greater than 3 months.
* Tumors with at least one of the following known mutations in the PI-3K signaling pathway, via assays performed in a CLIA-approved setting (Foundation Medicine FoundationOne test will be used. This assay uses a cut-off of 5% allele fraction for mutations. Allele fraction will be requested on each sample):

  1. PIK3CA,
  2. PIK3CG,
  3. PIK3R1, PIK3R5 and PIK3AP1 (regulatory subunits),
  4. AKT and mTOR, or
  5. PTEN Note: PIK3CA amplification is not eligible.
* Prior receipt of platinum-containing chemotherapy for recurrent/metastatic disease or a history of progression of disease within 6 months of receiving platinum as part of concurrent chemoradiation.
* Disease must not be amenable to potentially curative treatment..
* Has recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy.

  * Myelosuppressive chemotherapy: At least 3 weeks since completion (6 weeks for nitrosourea)
  * Biologic (anti-neoplastic agent): At least 14 days since completion of therapy with a biologic agent.
  * Radiation (XRT):1 week must have elapsed from prior palliative XRT to non-target lesions.
* Adequate Bone Marrow Function Defined for all subjects (including status post SCT):

  * Peripheral absolute neutrophil count (ANC) 1000/mm3; Note: must be >7 days from use of hematopoietic growth factor or 21 days from pegfilgastrim
  * Platelet count 75,000/ mm3 (transfusion independent for >7 days)
  * Hemoglobin 8.0 g/dL (may receive transfusions)
* Adequate Renal Function Defined As:

  * Serum creatinine ≤ 1.5 x institution's ULN (upper limit of normal), or
  * Creatinine clearance 50 ml/min
* Adequate Liver and Pancreatic Function Defined As:

  * Total bilirubin 1.5 x upper limit of normal, and
  * ALT or AST 5 x upper limit of normal, and
  * Albumin 2 g/dL
* Adequate Central Nervous System Function Defined As:

  * Subjects with seizure disorder may be enrolled if on anticonvulsants and seizures are well controlled.

Exclusion Criteria:

* Brain metastases or spinal cord compression, unless treatment was completed at least 4 weeks before study entry, and stable without steroid treatment for at least 4 weeks.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac [including life threatening arrhythmias], hepatic, or renal disease).
* Unresolved toxicity ≥ CTCAE Grade 2 from previous anti-cancer therapy except alopecia or long-term radiation toxicity (radiation related toxicity 3 months or greater after radiation exposure).
* Presence of cardiac impairment defined as:

  * Prior history of cardiovascular disease including heart failure that meets New York Hearth Association (NYHA) class III and IV definitions; OR
  * History of myocardial infarction/active ischemic heart disease within one year of study entry; OR
  * Uncontrolled dysrhythmias; OR
  * Poorly controlled angina.
* Participation in a trial of an investigational agent within the prior 30 days.
* Pregnant or breast-feeding females.
* History of other malignancies except curatively excised carcinoma in situ of the cervix, non-melanomatous skin carcinoma or superficial bladder cancer or other solid tumors curatively treated with no evidence of disease for 3 years. Other cases will be reviewed and possibly allowed if discussed with and approved by the Principal Investigator.
* Patients receiving therapeutic doses of warfarin.
* Blood pressure greater than 170/90 or two standard deviations from normal based on age and weight nomogram on three separate measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SF1126
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | SF1126
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: To Determine ORR
Description: best response of PR or CR observed within 6 months of enrollment
Time Frame: 6 months
Arm/Group | SF1126
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Groups:
- SF1126: SF1126 1110 mg/m2 administered intravenously (IV) twice per week (separated by at least three days) for the first four treatment cycles (28 days) and then once weekly for subsequent cycles.
  SF1126
Arm/Group | SF1126
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: To Assess the Effect of SF1126 on Time to Progression.
Time Frame: 4 years
Arm/Group | SF1126
Number analyzed (Participants) | 0

4. Secondary Outcome: To Assess the Effect of SF1126 on Overall Survival.
Time Frame: 4 years
Arm/Group | SF1126
Number analyzed (Participants) | 0

5. Secondary Outcome: To Assess Disease-related Patient-reported Outcomes Using the EORTC-QLQ-
Time Frame: 4 years
Arm/Group | SF1126
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | SF1126
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SF1126 (N=1)
dyspnea (Cardiac disorders) | 1 (1)
atrial fibrilation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SF1126 (N=1)
anemia (Blood and lymphatic system disorders) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cardiac troponin T increased (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes